CLINICAL TRIAL: NCT05556421
Title: Can Uterocervical Angle Predict the Displacement of Copper Intrauterine Devices (T-Cu 380A)
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KanuniSSEAH2
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2022-09

CONDITIONS: Intrauterine Device
Keywords: displacement; contraception; family planning; T-Cu 380A; uterocervical angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- case group: dislocated intrauterine device
  Interventions: Diagnostic Test: uterocervical angle
- control group: normal intrauterine device position
  Interventions: Diagnostic Test: uterocervical angle

INTERVENTIONS:
Diagnostic Test: uterocervical angle — uterocervical angles were measured for both groups by transvaginal ultrasonography and investigated whether the uterocervical angle had any effect in predicting the displacement of copper intrauterine devices.

SUMMARY:
The investigators conducted a case-control study between December 2020-June 2021 at Istanbul Health Sciences University Kanuni Sultan Suleyman Training and Research Hospital family planning outpatient clinics. One hundred and forty-three patients who had copper intrauterine devices (T Cu 380 A) inserted for contraception were evaluated between the 6th week to 5 years after insertion. Patients were divided into two groups according to their ultrasonographic examinations as "displaced" or "normal" positions. Uterocervical angles were measured of both groups by transvaginal ultrasonography and investigated whether the uterocervical angle had any effect in predicting the displacement of copper intrauterine devices.

DETAILED DESCRIPTION:
Family planning contains various protection methods, and copper intrauterine devices (IUD) are one of these. It has come forward among the contraception methods due to its long-acting effect, rapid return of fertility when discontinued, and ease of use. In worldwide usage, IUDs are the third most common method of contraception after tubal ligation and male condoms (1). When long-acting contraception methods were compared, the failure rate of the IUD was 0.8% per 100 women within one year (2). Factors affecting failure were; the application time of IUDs (3), application technique (4), uterus dimensions (5), endometrial cavity length (6), parity (7), and mode of delivery (8).

Uterocervical angle (UCA) is the angle measured in the triangle region between the anterior uterine segment and the cervical canal (9). UCA has been evaluated to predict the threat of preterm birth in national and international studies (9,10). In the literature, UCA has not been used in any studies within the scope of family planning. Our study aimed to investigate the feasibility of uterocervical angle measurements in predicting the dislocation of IUDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 21-45

Exclusion Criteria:

1. Patients under the age of twenty-one and over the age of 45
2. Patients applied to the hospital within the first 6 weeks after copper IUD insertion
3. Patients with Space-occupying lesions (polyp, fibroid) in the uterine cavity
4. Patients who have and/or had a pelvic inflammatory disease
5. Patients who had Ascus, Hgsil, Lgsil, CIN (1,2,3), carcinoma in situ, and malignancy in their smear results before the study started or detected during the study period, and patients who were done LEEP or conization procedures due to these pathologies.
6. Patients with Descensus uteri
7. Patients with cervical polyps
8. Patients with connective tissue disease I- Patients with uterine myomas or adenomyosis
9. Patients with uterine anomaly
10. Patients with vaginal infection or recurrent vaginitis and patients with abnormal uterine bleeding

l- Patients with immune-compromised situations such as AIDS, drug use, or cortisone treatment m- Patients using anticoagulants for any reason n- Patients who have known Copper allergy or rare Copper metabolism disease (Wilson disease)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The female patients between the ages of 21-45 who applied to either gynecology or family planning outpatient clinics and who had been using copper IUD (T Cu 380-A) as a contraception method for the last 6 weeks to 5 years were included in the study. Patients were included in the study on a voluntary basis.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
uterocervical angle | 6 months
  Uterocervical angle (UCA) is the angle measured in the triangle region between the anterior uterine segment and the cervical canal

SECONDARY OUTCOMES:
uterine volume | 6 months
  Uterine volume was accepted as ellipsoid with transvaginal ultrasonography device measured in transverse, longitudinal, and antero-posterior planes and volume was calculated in cm3.
endometrial cavity length | 6 months
  The length of the endometrial cavity (ECL) was determined as the canal extending from the beginning of the internal cervical os to the uterine fundus endometrium.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No